CLINICAL TRIAL: NCT02093884
Title: Texting 2 Initiate: A Pilot Study Using Text Messaging to Communicate With Adolescent Females in the Pediatric Emergency Department (T2I)
Brief Title: A Pilot Study Using Text Messaging to Communicate With Adolescent Females in the Pediatric Emergency Department
Acronym: T2I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Lauren S. Chernick, Assistant Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAM3457
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; Pregnancy, unplanned; Reproductive behavior; Pregnancy in Adolescence; Text messaging
MeSH Terms: conditions — Reproductive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Messaging Intervention (Experimental): Patients in the text messaging group will receive educational and motivational text messages.
  Interventions: Other: Text Messaging Intervention
- Standard Referral (Active Comparator): Patients in the standard referral arm will receive paper based information about the Family Planning Clinic.
  Interventions: Other: Standard Referral

INTERVENTIONS:
Other: Text Messaging Intervention
  Arms: Text Messaging Intervention
Other: Standard Referral
  Arms: Standard Referral

SUMMARY:
The objective of this study is to develop and test an emergency department (ED)-based intervention which uses text messages to facilitate contraception initiation.

DETAILED DESCRIPTION:
Our hypothesis is that adolescent females at high pregnancy risk who receive text message reminders and motivational messages that promote contraception and referral to the Family Planning Clinic are more likely to start effective contraception than those who receive standard paper-based referral to the Family Planning Clinic alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-19 years
* Sexually active with males in the past three months
* Presenting to the ED for a reproductive health complaint.

Exclusion Criteria:

* Presently pregnant
* Too ill for participation per the attending physician
* Cognitively impaired
* In foster care or a ward of the state
* Does not speak English or Spanish
* Does not own a cellular or mobile phone with text messaging capabilities
* Used contraception at last intercourse and/or is currently using any "highly effective" or "effective" form of contraception (as defined by the World Health Organization)
* Does not live in Manhattan or the Bronx

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Initiation of highly effective contraception, as defined by the World Health Organization. | 3 months after initial enrollment
  We will be assessing contraception initiation rates based on electronic medical record review and telephone call follow up.

SECONDARY OUTCOMES:
Patient visits to Family Planning Clinic | 3 months after initial enrollment
  We assess Family Planning Clinic visits using our electronic medical records.
Follow up for contraceptive counseling to a doctor or nurse | 3 months after initial enrollment
  We will be asking patients during our phone call follow if they have had contraceptive counseling with any healthcare professional. We will also be looking through electronic medical records for documentation of contraceptive counseling such as by ICD-9 coding or a physician's/nurse's note.
Change in pregnancy intentions | 3 months after initial enrollment
  We will compare pregnancy intentions elicited from the answers provided in the baseline questionnaire to those reported on the telephone follow up for both study arms.

OTHER OUTCOMES:
Text messaging intervention safety | 3 months after initial enrollment
  Safety will be assessed during the telephone follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Chernick, MD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital Emergency Department, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730